CLINICAL TRIAL: NCT02226835
Title: An Investigation of Retinal Findings in Patients With Signs and Symptoms of Alzheimer's Disease Enrolled in 09-M-0198
Brief Title: Study of Retinal Findings in People With Signs and Symptoms of Alzheimer s Disease Enrolled in 09-M-0198
Status: Terminated | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 140173; 14-EI-0173
Record Dates: First submitted 2014-08-26; First posted 2014-08-27 (Estimated); Last update posted 2018-09-27 (Actual); Status verified 2017-01-24

CONDITIONS: Age-Related Macular Degeneration; Alzheiner's Disease; AMD
Keywords: OCT; Alzheimer's Disease; Age-Related Macular Degeneration (AMD)
MeSH Terms: conditions — Macular Degeneration; Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
Background:

- Alzheimer s disease affects the brain and causes memory and thinking problems in older people. Macular degeneration (MD) is an eye condition. It is the leading reason that people over age 55 in the United States lose their central vision. Central vision is important for seeing fine details and for tasks like reading and driving. A feature of Alzheimer s disease is plaques in the brain. A feature of age-related MD is deposits in the retina in the eye. Researchers want to learn more about these diseases and find out if they are related.

Objective:

- To see whether there is a relationship between Alzheimer s disease and age-related macular degeneration.

Eligibility:

- People with or without Alzheimer s disease enrolled in another study. Participants must have someone to help them take part in this study.

Design:

* Participants will be screened through the other study. They will have 1 visit. The tests will take about 3 hours.
* Participants will answer questions about their medical and eye history.
* Participants will have an eye exam to test how well they see. Their eye pressure will be measured and their eye movements will be checked.
* Participants will get eye drops to dilate their pupils. Researchers will take pictures of the retina and the inside of the eye. Researchers may measure the thickness of the retina.
* Participants will continue to receive care from their regular eye doctor during and after the study.

DETAILED DESCRIPTION:
Objective:

Age-related macular degeneration (AMD) and Alzheimer s disease (AD) are both neurodegenerative diseases which affect a similar demographic of patients. Beyond age being a common risk factor for both diseases, an important common characteristic is a similarity in pathology findings, specifically, the presence of amyloid (beta) (A(beta)) in the senile plaques of the AD brain and in the drusen of AMD patients. As both of these diseases are the cause of significant morbidity of the quickly growing aging population, understanding the pathogenesis of both and identification of any overlapping pathophysiology will lead to a better understanding of each disease. The objective of this study is to investigate the presence of AMD and other neurodegenerative lesions and characterize retinal findings in a group of participants with well-phenotyped AD.

Study Population:

Up to 150 participants (100 symptomatic, 50 controls) will be recruited from patients already enrolled and participating in the National Institute of Mental Health (NIMH) study, 09-M-0198, Screening and Evaluation of Patients with Signs and Symptoms of Alzheimer s Disease.

Design:

This is a single center, cross-sectional, observational study that will include a single eye clinic visit with eye exam, visual acuity, photography and optical coherence tomography (OCT) testing.

Outcome Measures:

The primary outcome is the presence of AMD or other retinal findings in patients diagnosed with AD. Secondary outcomes will include autofluorescence imaging, spectral domain OCT and visual acuity.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patient must be enrolled in the 09-M-0198 protocol.
* In those participants that require special assistance, we will request that they be accompanied by a care taker to provide proper care and monitoring.

EXCLUSION CRITERIA:

Patients:

* The diagnosis of a different type of dementia, including frontotemporal dementia, normal pressure hydrocephalus, Lewy body dementia, Parkinson s disease dementia, Huntington s disease, or vascular dementia.
* Any medical contraindication to the procedures performed in the study, or any current severe medical or psychiatric illness other than Alzheimer s disease.
* Behavioral symptoms that would preclude the gathering of data for the study, or advanced disease such that participants cannot provide assent.

Controls:

* The diagnosis of a brain disorder.
* Any medical contraindication to the procedures performed in the study, or any current severe medical or psychiatric illness.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-08-13; Primary Completion 2017-01-24 (Actual); Study Completion 2017-01-24 (Actual)

PRIMARY OUTCOMES:
Photographs and images of subjects' eyes | Study completion

SECONDARY OUTCOMES:
OCT measurement | Study completion

CONTACTS AND LOCATIONS:
Overall Officials: Catherine A Cukras, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Friedman DS, O'Colmain BJ, Munoz B, Tomany SC, McCarty C, de Jong PT, Nemesure B, Mitchell P, Kempen J; Eye Diseases Prevalence Research Group. Prevalence of age-related macular degeneration in the United States. Arch Ophthalmol. 2004 Apr;122(4):564-72. doi: 10.1001/archopht.122.4.564. PMID 15078675
- [Background] Ferris FL 3rd, Fine SL, Hyman L. Age-related macular degeneration and blindness due to neovascular maculopathy. Arch Ophthalmol. 1984 Nov;102(11):1640-2. doi: 10.1001/archopht.1984.01040031330019. PMID 6208888
- [Background] Hebert LE, Scherr PA, Bienias JL, Bennett DA, Evans DA. Alzheimer disease in the US population: prevalence estimates using the 2000 census. Arch Neurol. 2003 Aug;60(8):1119-22. doi: 10.1001/archneur.60.8.1119. PMID 12925369